CLINICAL TRIAL: NCT05530122
Title: The Long-term Outcome of Patients With Ulcerative Colitis Treated With First Trial of Biological.
Brief Title: Prognosis in UC After First Biological
Acronym: biological
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Heli T Eronen, Principal investigator, Tampere University Hospital
Other Study IDs: R20543
Record Dates: First submitted 2022-08-29; First posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Ulcerative Colitis
Keywords: infliximab; adalimumab; golimumab; ustekinumab; vedolizumab; tofacitinib
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Infliximab; Adalimumab; golimumab; vedolizumab; Ustekinumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: infliximab, adalimumab, golimumab, vedolizumab, ustekinumab
  Other Names: small molecules

SUMMARY:
To study the long-term clinical outcome of patients with ulcerative colitis treated with first trial of biological therapy.

DETAILED DESCRIPTION:
UC patients treated with at least one biological in Tampere University Hospital between January 2009 and January 2020 were identified and reviewed from patient records.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated for ulcerative colitis for the first trial of biological

Exclusion Criteria:

* Age under 16 years

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients treated in Tampere University Hospital for UC between January 2009 and January 2020 were identified from the digital patient records. Patients at the age of 16 years or over with biological treatment initiated for treatment of moderate to severe UC were included.
Sampling Method: Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
Response to treatment | within 5 years
  Need for colectomy or enhancement of treatment within follow-up
Side-effects | within 5 years
  treatment related side-effects reported

CONTACTS AND LOCATIONS:
Overall Officials: Pekka Collin, PhD, Study Director — Tampere University Hospital; Heli Eronen, Principal Investigator — Central Hospital of Kanta-Häme

IPD SHARING:
Plan to Share IPD: No